CLINICAL TRIAL: NCT02890381
Title: Phase I Placebo-Controlled Study of the Infectivity, Safety and Immunogenicity of a Single Dose of a Recombinant Live-Attenuated Respiratory Syncytial Virus Vaccine, LID cp ΔM2-2, Lot RSV#009B, Delivered as Nose Drops to RSV-Seronegative Infants 6 to 24 Months of Age
Brief Title: Evaluating the Infectivity, Safety and Immunogenicity of a Recombinant Live-Attenuated Respiratory Syncytial Virus Vaccine (RSV LID cp ΔM2-2) in RSV-Seronegative Infants 6 to 24 Months of Age
Acronym: LID
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Interim data indicated this vaccine will not meet the protocol criteria for a good vaccine candidate.
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IMPAACT 2012; 30073 (Registry Identifier: DAIDS-ES Registry Number)
Record Dates: First submitted 2016-08-31; First posted 2016-09-07 (Estimated); Results first posted 2018-07-02 (Actual); Last update posted 2021-11-05 (Actual); Status verified 2018-05

CONDITIONS: Respiratory Syncytial Virus Infections
MeSH Terms: conditions — Respiratory Syncytial Virus Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- RSV LID cp ΔM2-2 Vaccine (Experimental): Participants received a single dose of the RSV LID cp ΔM2-2 vaccine at study entry (Day 0).
  Interventions: Biological: RSV LID cp ΔM2-2 Vaccine
- Placebo (Placebo Comparator): Participants received a single dose of placebo at study entry (Day 0).
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: RSV LID cp ΔM2-2 Vaccine — 10^5 plaque-forming units (PFUs); administered as nose drops
  Arms: RSV LID cp ΔM2-2 Vaccine
Biological: Placebo — Isotonic diluent, administered as nose drops
  Arms: Placebo

SUMMARY:
The purpose of this study was to evaluate the safety, infectivity, and immunogenicity of a single intranasal dose of a recombinant live-attenuated respiratory syncytial virus (RSV) vaccine in RSV-seronegative infants 6 to 24 months of age.

This study was a companion study to CIR 312.

DETAILED DESCRIPTION:
Human respiratory syncytial virus (RSV) is the most common viral cause of serious acute lower respiratory illness (LRI) in infants and children under 5 years of age worldwide. This study evaluated the safety, infectivity, and immunogenicity of a single dose of RSV LID cp ΔM2-2, a recombinant live-attenuated RSV vaccine, in RSV-seronegative infants 6 to 24 months of age.

Participants were randomly assigned to receive a single dose of the RSV LID cp ΔM2-2 vaccine or placebo at study entry (Day 0).

Participants were enrolled in the study between April 1 and October 14 (outside of RSV season) and remained on study until they completed the post-RSV season visit between April 1 and April 30 in the calendar year following enrollment. Participants' total study duration was between 6 and 10 months, depending on when they enrolled in the study. Participants attended several study visits throughout the study, which may include physical examinations, blood collection, and nasal washes. Participants' parents or guardians were contacted by study staff at various times during the study to monitor participants' health.

The study was closed to accrual early after interim data were reviewed by a subset of protocol team members and it was concluded that this vaccine candidate will not meet the criteria listed in the protocol for a good vaccine candidate. This recommendation was shared with the (blinded) protocol chair and the Medical Officers, as well as the Data Safety and Monitoring Board (DSMB), who agreed with the unblinded protocol team members' assessment. The targeted sample size was 33 (22 in the vaccine arm and 11 in the placebo arm). Participants already on study at the time of the early closing decision remained on study and completed the follow-up per protocol.

ELIGIBILITY:
Inclusion Criteria:

* Greater than or equal to 6 months (defined as greater than or equal to 180 days) of age at the time of screening and less than 25 months (defined as less than 750 days) of age.
* Good health based on review of the medical record, history, and physical examination, without evidence of chronic disease.
* Parents/guardians willing and able to provide written informed consent as described in the protocol.
* Seronegative for RSV antibody, defined as a serum RSV-neutralizing antibody titer less than 1:40 at screening from a sample collected no more than 42 days prior to inoculation. Note: results from specimens collected during screening for IMPAACT 2011 were acceptable as long as within the 42-day window.
* Growing at a normal velocity for age (as demonstrated on a standard growth chart) AND

  * If less than 1 year of age: current height and weight above the 5th percentile.
  * If 1 year of age or older: current height and weight above the 3rd percentile for age.
* Received routine immunizations appropriate for age (as per national Center for Disease Control Advisory Committee on Immunization Practices [ACIP]).
* Expected to be available for the duration of the study.
* If born to an HIV-infected woman, participant must not have been breastfed and must have had documentation of 2 negative HIV nucleic acid (RNA or DNA) test results from samples collected on different dates with both collected when greater than or equal to 1 month of age and at least one collected when greater than or equal to 4 months of age, and no positive HIV nucleic acid (RNA or DNA) test; or 2 negative HIV antibody tests, both from samples collected at greater than or equal to 6 months of age.

Exclusion Criteria:

* Known or suspected HIV infection or impairment of immunological functions.
* Receipt of immunosuppressive therapy, including any systemic, including either nasal or inhaled, corticosteroids within 28 days of enrollment. Note: Cutaneous (topical) steroid treatment is not an exclusion.
* Bone marrow/solid organ transplant recipient.
* Major congenital malformations (such as congenital cleft palate) or cytogenetic abnormalities.
* Previous receipt of a licensed or investigational RSV vaccine (or placebo in any IMPAACT RSV study) or previous receipt of or planned administration of any anti-RSV product (such as ribavirin or RSV IG or RSV mAb).
* Previous anaphylactic reaction.
* Previous vaccine-associated adverse reaction that was Grade 3 or above.
* Known hypersensitivity to any study product component.
* Heart disease. Note: Participants with cardiac abnormalities documented to be clinically insignificant and requiring no treatment were allowed to enroll.
* Lung disease, including any history of reactive airway disease or medically documented wheezing.
* Member of a household that contains, or will contain, an infant who is less than 6 months of age at the enrollment date through Day 28.
* Member of a household that contains another child enrolled, or scheduled to be enrolled in IMPAACT 2011, 2012 or 2013 AND an overlap in residency during that other child's participation in the study's Acute Phase (Days 0 to 28).
* Member of a household that contains an immunocompromised individual, including, but not limited to:

  * a person who is greater than or equal to 6 years of age with HIV-related immunodeficiency, defined as having a most recent CD4 T lymphocyte cell count less than 300 cells/mm^3. CD4 T lymphocyte count must have been measured within 6 months prior to enrollment, or
  * a person age 1 year up to less than 6 years with HIV-related immunodeficiency, defined as having a most recent CD4 T lymphocyte cell percentage less than 25 or CD4 T lymphocyte count less than 750 cells/mm^3 (if both values available, use the lower of the two). CD4 T lymphocyte parameter must have been measured within the 6 months prior to enrollment; or
  * a person age less than 1 year with HIV-related immunodeficiency, defined as having a most recent CD4 T lymphocyte cell percentage less than 30 or CD4 T lymphocyte count less than 1000 cells/mm^3 (if both values available, use the lower of the two). CD4 T lymphocyte parameter must have been measured within the 6 months prior to enrollment; or
  * a person who has received chemotherapy within the 12 months prior to enrollment; or
  * a person receiving immunosuppressant agents; or
  * a person living with a solid organ or bone marrow transplant.

Verbal report of CD4 T cell lymphocyte is sufficient documentation if the parent/guardian is confident of history.

* Attends a daycare facility and shares a room with infants less than 6 months of age, and parent/guardian is unable or unwilling to suspend daycare for 28 days following inoculation.
* Any of the following events at the time of enrollment:

  * fever (rectal temperature of greater than or equal to 100.4°F (38°C)), or
  * upper respiratory signs or symptoms (rhinorrhea, cough, or pharyngitis) or
  * nasal congestion significant enough to interfere with successful inoculation, or
  * otitis media.
* Receipt of the following prior to enrollment:

  * any killed vaccine or live-attenuated rotavirus vaccine within the 14 days prior, or
  * any live vaccine, other than rotavirus vaccine, within the 28 days prior, or
  * another investigational vaccine or investigational drug within 28 days prior
* Scheduled administration of the following after planned inoculation:

  * killed vaccine or live-attenuated rotavirus vaccine within the 14 days after, or
  * any live vaccine other than rotavirus in the 28 days after, or
  * another investigational vaccine or investigational drug in the 56 days after
* Receipt of immunoglobulin, any antibody products, or any blood products within the past 6 months.
* Receipt of any of the following medications within 3 days of study enrollment:

  * systemic antibacterial, antiviral, antifungal, anti-parasitic, or antituberculous agents, whether for treatment or prophylaxis, or
  * intranasal medications, or
  * other prescription medication except as listed below

Permitted concomitant medications (prescription or non-prescription) include nutritional supplements, medications for gastroesophageal reflux, eye drops, and topical medications, including (but not limited to) cutaneous (topical) steroids, topical antibiotics, and topical antifungal agents.

* Receipt of salicylate (aspirin) or salicylate-containing products within the 28 days prior to enrollment.
* Born at less than 34 weeks gestation.
* Born at less than 37 weeks gestation and less than 1 year of age at the time of enrollment.
* Suspected or documented developmental disorder, delay, or other developmental problem.
* Previous receipt of supplemental oxygen therapy in a home setting.

Ages: 6 Months to 24 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 17 (Actual)
Dates: Start 2016-10-05 (Actual); Primary Completion 2017-04-24 (Actual); Study Completion 2017-04-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Coleen Cunningham, MD, Study Chair — Children's Health Center, DUMC
Locations (5):
- United States (5):
  - David Geffen School of Medicine at UCLA NICHD CRS, Los Angeles, California
  - Univ. of Colorado Denver NICHD CRS, Aurora, Colorado
  - Rush Univ. Cook County Hosp. Chicago NICHD CRS, Chicago, Illinois
  - Johns Hopkins University Center for Immunization Research, Baltimore, Maryland
  - Philadelphia IMPAACT Unit CRS, Philadelphia, Pennsylvania

REFERENCES:
- [Derived] Cunningham CK, Karron R, Muresan P, McFarland EJ, Perlowski C, Libous J, Thumar B, Gnanashanmugam D, Moye J Jr, Schappell E, Barr E, Rexroad V, Aziz M, Deville J, Rutstein R, Yang L, Luongo C, Collins P, Buchholz U; International Maternal Pediatric Adolescent AIDS Clinical Trials (IMPAACT) 2012 Study Team. Live-Attenuated Respiratory Syncytial Virus Vaccine With Deletion of RNA Synthesis Regulatory Protein M2-2 and Cold Passage Mutations Is Overattenuated. Open Forum Infect Dis. 2019 May 6;6(6):ofz212. doi: 10.1093/ofid/ofz212. eCollection 2019 Jun. PMID 31211158
- See also: DAIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table), Version 2.0, November 2014 — http://rsc.tech-res.com/docs/default-source/safety/daids_ae_grading_table_v2_nov2014.pdf?sfvrsn=8
- See also: Description: Manual for Expedited Reporting of Adverse Events to DAIDS (DAIDS EAE Manual), Version 2.0, January 2010 — http://rsc.tech-res.com/docs/default-source/safety/manual_for_expedited_reporting_aes_to_daids_v2.pdf?sfvrsn=12

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period was from September to October 2016. Participants were recruited from medical clinics.
Groups:
- Placebo: Participants received a single dose of placebo at study entry (Day 0).
  Placebo: Administered as nose drops
Period: Overall Study
Arm/Group | RSV LID cp ΔM2-2 Vaccine | Placebo
Started | 11 | 6
Completed | 11 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Analysis population was all participants enrolled.
Groups:
- Total: Total of all reporting groups
Arm/Group | RSV LID cp ΔM2-2 Vaccine | Placebo | Total
Number analyzed (Participants) | 11 | 6 | 17
Age, Continuous [Median (Inter-Quartile Range); unit: months] | 12 [8 to 15] | 9 [6 to 12] | 10 [8 to 14]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 10
  Male | 5 | 2 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 8 | 6 | 14
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 2 | 5
  White | 6 | 2 | 8
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 11 | 6 | 17
Serum RSV-neutralizing antibody titers [Median (Inter-Quartile Range); unit: log 2 titers] — Data values are presented as log 2 titers.
  log 2 titers | 2.3 [2.3 to 3.6] | 2.3 [2.3 to 3.7] | 2.3 [2.3 to 3.6]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Solicited Adverse Events (AEs) by Grade
Description: Solicited adverse events include fever; otitis media; upper respiratory illness (URI); lower respiratory illness (LRI) and cough (without LRI). The number of participants who experienced solicited adverse events was presented. A participant was only counted once in each solicited AE category, and that is in the line corresponding to the highest grade adverse event they had in that category. These events were graded (Grade 1-mild to Grade 4-life-threatening) following protocol-defined grading system outlined in Table 3 and Table 4 in the protocol document.
Time Frame: Measured from Day 0 through Day 28
Population: All study participants were included.
Measure: Count of Participants; unit: Participants
Arm/Group | RSV LID cp ΔM2-2 Vaccine | Placebo
Number analyzed (Participants) | 11 | 6
Participants
  Fever: Did not have this AE | 9 | 2
  Fever: Grade 1 | 0 | 2
  Fever: Grade 2 | 1 | 1
  Fever: Grade 3 | 1 | 1
  Fever: Grade 4 | 0 | 0
  Otitis Media: Did not have this AE | 8 | 6
  Otitis Media: Grade 1 | 0 | 0
  Otitis Media: Grade 2 | 3 | 0
  Otitis Media: Grade 3 | 0 | 0
  Otitis Media: Grade 4 | 0 | 0
  Upper Respiratory Illness (URI): Did not have this AE | 5 | 0
  Upper Respiratory Illness (URI): Grade 1 | 6 | 6
  Upper Respiratory Illness (URI): Grade 2 | 0 | 0
  Upper Respiratory Illness (URI): Grade 3 | 0 | 0
  Upper Respiratory Illness (URI): Grade 4 | 0 | 0
  Lower Respiratory Illness (LRI) with RSV shedding: Did not have this AE | 11 | 6
  Lower Respiratory Illness (LRI) with RSV shedding: Grade 1 | 0 | 0
  Lower Respiratory Illness (LRI) with RSV shedding: Grade 2 | 0 | 0
  Lower Respiratory Illness (LRI) with RSV shedding: Grade 3 | 0 | 0
  Lower Respiratory Illness (LRI) with RSV shedding: Grade 4 | 0 | 0
  LRI in the absence of RSV shedding: Did not have this AE | 9 | 6
  LRI in the absence of RSV shedding: Grade 1 | 0 | 0
  LRI in the absence of RSV shedding: Grade 2 | 2 | 0
  LRI in the absence of RSV shedding: Grade 3 | 0 | 0
  LRI in the absence of RSV shedding: Grade 4 | 0 | 0
  Cough, without LRI: Did not have this AE | 7 | 2
  Cough, without LRI: Grade 1 | 4 | 4
  Cough, without LRI: Grade 2 | 0 | 0
  Cough, without LRI: Grade 3 | 0 | 0
  Cough, without LRI: Grade 4 | 0 | 0
Statistical Analysis 1: Comparison: RSV LID cp ΔM2-2 Vaccine; Test type: Other; % vaccine recipients with solicited AEs = 64, 90% CI 2-sided [35 to 86]
Statistical Analysis 2: Comparison: Placebo; Test type: Other; % placebo recipients with solicited AEs = 100, 90% CI 2-sided [61 to 100]

2. Primary Outcome: Number of Participants With Unsolicited AEs by Grade
Description: Unsolicited adverse events were other events, not included in the solicited AEs. The number of participants who experienced solicited adverse events was presented. A participant was only counted once in each unsolicited AE category, and that is in the line corresponding to the highest grade adverse event they had in that category. AE grading (Grade 1- mild to Grade 4-life-threatening) was done by DAIDS AE Grading table v2.0 (see References).
Time Frame: Measured from Day 0 through Day 28
Population: All participants were included.
Measure: Count of Participants; unit: Participants
Arm/Group | RSV LID cp ΔM2-2 Vaccine | Placebo
Number analyzed (Participants) | 11 | 6
Participants
  Nasal Congestion: No adverse event | 9 | 4
  Nasal Congestion: Grade 1 | 2 | 2
  Nasal Congestion: Grade 2 | 0 | 0
  Nasal Congestion: Grade 3 | 0 | 0
  Nasal Congestion: Grade 4 | 0 | 0
  Discomfort: No adverse event | 10 | 4
  Discomfort: Grade 1 | 1 | 2
  Discomfort: Grade 2 | 0 | 0
  Discomfort: Grade 3 | 0 | 0
  Discomfort: Grade 4 | 0 | 0
  Vomiting, Diarrhea, Constipation: No adverse event | 9 | 5
  Vomiting, Diarrhea, Constipation: Grade 1 | 2 | 1
  Vomiting, Diarrhea, Constipation: Grade 2 | 0 | 0
  Vomiting, Diarrhea, Constipation: Grade 3 | 0 | 0
  Vomiting, Diarrhea, Constipation: Grade 4 | 0 | 0
  Eczema: No adverse event | 11 | 5
  Eczema: Grade 1 | 0 | 1
  Eczema: Grade 2 | 0 | 0
  Eczema: Grade 3 | 0 | 0
  Eczema: Grade 4 | 0 | 0
  Conjunctivitis: No adverse event | 10 | 6
  Conjunctivitis: Grade 1 | 0 | 0
  Conjunctivitis: Grade 2 | 1 | 0
  Conjunctivitis: Grade 3 | 0 | 0
  Conjunctivitis: Grade 4 | 0 | 0
  Irritability: No adverse event | 10 | 6
  Irritability: Grade 1 | 1 | 0
  Irritability: Grade 2 | 0 | 0
  Irritability: Grade 3 | 0 | 0
  Irritability: Grade 4 | 0 | 0
Statistical Analysis 1: Comparison: RSV LID cp ΔM2-2 Vaccine; Test type: Other; % vaccinees with unsolicited AEs = 36, 90% CI 2-sided [14 to 65]
Statistical Analysis 2: Comparison: Placebo; Test type: Other; % placebo with unsolicited AEs = 50, 90% CI 2-sided [15 to 85]

3. Primary Outcome: Number of Participants With Serious Adverse Events (SAEs)
Description: A Serious Adverse Event (SAE) is an AE, whether considered related to the study product or not, that:
  1. Results in death during the period of protocol-defined surveillance
  2. Is life threatening: defined as an event in which the patient was at immediate risk of death at the time of the event; it does not refer to an event that hypothetically might have caused death were it more severe
  3. Requires inpatient hospitalization (or prolongation of existing hospitalization): defined as at least an overnight stay in the hospital or emergency ward for treatment that would have been inappropriate if administered in the outpatient setting
  4. Results in a persistent or significant disability/incapacity
  5. Is a congenital anomaly or birth defect
  6. Is an important medical event that may not be immediately life threatening or result in death or hospitalization but may jeopardize the patient or may require intervention to prevent one of the outcomes listed above.
Time Frame: Measured from Day 0 through Day 56
Population: All participants were included.
Measure: Count of Participants; unit: Participants
Arm/Group | RSV LID cp ΔM2-2 Vaccine | Placebo
Number analyzed (Participants) | 11 | 6
Participants | 0 | 0

4. Primary Outcome: Number of Participants Infected With RSV Vaccine
Description: Defined as 1) vaccine virus identified in a nasal wash from Study Day 0-28 (a binary outcome based on nasal washes) or 2) greater than or equal to 4-fold rise in serum RSV-neutralizing antibody titer between Study Days 0 and 56.
Time Frame: Measured at Days 0, 3, 5, 7, 10, 12, 14, 17, and 28 for nasal washes, and at Days 0, 56 for serum RSV-neutralizing antibodies
Population: All participants were included.
Measure: Count of Participants; unit: Participants
Arm/Group | RSV LID cp ΔM2-2 Vaccine | Placebo
Number analyzed (Participants) | 11 | 6
Participants | 6 | 0

5. Primary Outcome: Peak Titer of Vaccine Virus Shed
Description: This is the highest value per participant of the titer of vaccine virus shed. It was measured by culture. Only participants who met the definition of infection with vaccine virus were included.
Time Frame: Measured at Days 0, 3, 5, 7, 10, 12, 14, 17, and 28
Population: Only participants who met the definition of infection with vaccine virus were included.
Measure: Median (Inter-Quartile Range); unit: log 10 Plaque Forming Units (PFU)/mL
Arm/Group | RSV LID cp ΔM2-2 Vaccine | Placebo
Number analyzed (Participants) | 6 | 0
log 10 Plaque Forming Units (PFU)/mL | 1.6 [0.5 to 3.4] |

6. Primary Outcome: Duration of Virus Shedding in Nasal Washes
Description: Determined separately by a) culture and b) reverse transcription polymerase chain reaction (RT-PCR)
Time Frame: Measured at Days 0, 3, 5, 7, 10, 12, 14, 17, and 28. Last day positive is reported.
Population: Only participants who met the definition of infection were included.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | RSV LID cp ΔM2-2 Vaccine | Placebo
Number analyzed (Participants) | 6 | 0
days
  Culture positive | 6 [0 to 12] |
  RT-PCR positive | 12 [0 to 15] |

7. Primary Outcome: Number of Participants With a Greater Than or Equal to 4-fold Rise in Serum RSV-neutralizing Antibody Titer
Description: Immunogenicity was assessed pre-inoculation, and at approximately 2 months post-inoculation (Study Day 56). Antibody responses were defined as a greater than or equal to 4-fold increase in titer in paired specimens, between pre and post time points.
Time Frame: Measured at Day 0 and Day 56
Population: One placebo recipient had missing data at the Day 56 evaluation. All other participants were included.
Measure: Count of Participants; unit: Participants
Arm/Group | RSV LID cp ΔM2-2 Vaccine | Placebo
Number analyzed (Participants) | 11 | 5
Participants | 5 | 2
Statistical Analysis 1: Comparison: RSV LID cp ΔM2-2 Vaccine vs Placebo; Test type: Superiority; p = 0.64, Fisher Exact — Since the sample sizes are unequal, at the suggestion of the DSMB statistician, a 1-sided Fisher's exact test was used to test the hypothesis that the proportions of >=4-fold rises were higher in the vaccinated group than in the placebo group

8. Primary Outcome: Serum Antibody Responses to RSV F Glycoprotein as Assessed by Enzyme-linked Immunosorbent Assay (ELISA)
Description: Immunogenicity was assessed at approximately 2 months post-inoculation (Study Day 56).
Time Frame: Measured at Day 56
Population: One placebo recipient had missing data at Day 56. All other participants were included.
Measure: Median (Inter-Quartile Range); unit: log 2 titers
Arm/Group | RSV LID cp ΔM2-2 Vaccine | Placebo
Number analyzed (Participants) | 11 | 5
log 2 titers | 12.3 [5.7 to 14.2] | 8.2 [7.1 to 15.2]
Statistical Analysis 1: Comparison: RSV LID cp ΔM2-2 Vaccine vs Placebo; Test type: Superiority; p = 0.73, Log Rank — The threshold for statistical significance is 0.05

9. Secondary Outcome: Number of Participants Who Had Symptomatic, Medically Attended Respiratory and Febrile Illness, by Grade, Among Those Who Experienced Natural Infection With wt RSV During the Subsequent RSV Season
Description: The number of participants who had symptomatic, medically attended respiratory and febrile illness among those who had RSV detected in nasal washes or >=4 fold rise in serum antibodies during the subsequent RSV season were presented. A participant was only counted once in each solicited AE category, and that was in the line corresponding to the highest grade adverse event they had in that category.
Time Frame: Measured through participant's last study visit, up to a total of 6 to 10 months depending on when participants enroll in the study
Population: Only participants who had RSV detected in nasal washes or >=4 fold rise in serum antibodies during the subsequent RSV season were included.
Measure: Count of Participants; unit: Participants
Arm/Group | RSV LID cp ΔM2-2 Vaccine | Placebo
Number analyzed (Participants) | 3 | 2
Participants
  Fever: No adverse event | 2 | 1
  Fever: Grade 1 | 1 | 1
  Fever: Grade 2 | 0 | 0
  Fever: Grade 3 | 0 | 0
  Fever: Grade 4 | 0 | 0
  Otitis Media: No adverse event | 1 | 2
  Otitis Media: Grade 1 | 1 | 0
  Otitis Media: Grade 2 | 1 | 0
  Otitis Media: Grade 3 | 0 | 0
  Otitis Media: Grade 4 | 0 | 0
  URI: No adverse event | 1 | 2
  URI: Grade 1 | 2 | 0
  URI: Grade 2 | 0 | 0
  URI: Grade 3 | 0 | 0
  URI: Grade 4 | 0 | 0
  LRI: No adverse event | 0 | 1
  LRI: Grade 1 | 0 | 0
  LRI: Grade 2 | 2 | 1
  LRI: Grade 3 | 1 | 0
  LRI: Grade 4 | 0 | 0
  Cough, without LRI: No adverse event | 0 | 1
  Cough, without LRI: Grade 1 | 1 | 0
  Cough, without LRI: Grade 2 | 2 | 1
  Cough, without LRI: Grade 3 | 0 | 0
  Cough, without LRI: Grade 4 | 0 | 0

10. Secondary Outcome: Magnitude of Serum RSV-neutralizing Antibody Responses in the Vaccine and Placebo Recipients Who Experience Natural Infection With wt RSV During the Subsequent RSV Season.
Description: Only participants who had RSV detected in nasal washes or a greater than or equal to 4-fold rise in serum antibodies during the subsequent RSV season were included. RSV-neutralizing antibody titers were measured pre- and post-RSV surveillance season.
Time Frame: as for outcome 9
Population: Only participants who had RSV detected in nasal washes or a greater than or equal to 4-fold rise in serum antibodies during the subsequent RSV season were included.
Measure: Median (Inter-Quartile Range); unit: log 2 titers
Arm/Group | RSV LID cp ΔM2-2 Vaccine | Placebo
Number analyzed (Participants) | 3 | 2
log 2 titers
  Pre RSV surveillance | 2.3 [2.3 to 3.9] | 2.3 [2.3 to 2.3]
  Post RSV Surveillance | 7.4 [6.5 to 11.0] | 6.9 [6.8 to 7.0]

11. Secondary Outcome: Number of Participants With B Cell Responses to Vaccine
Description: A B cell response to vaccine is indicated by a greater than or equal to 4-fold change in serum antibody titers to RSV F glycoprotein between the pre- and post-inoculation time points, and between pre- and post-RSV surveillance time points.
Time Frame: as for outcome 9
Population: One placebo recipient had missing data for the Day 56 and the pre-RSV surveillance time points. All other participants were included.
Measure: Count of Participants; unit: Participants
Arm/Group | RSV LID cp ΔM2-2 Vaccine | Placebo
Number analyzed (Participants) | 11 | 5
Participants
  From pre- to post-inoculation | 5 | 2
  From pre- to post-RSV surveillance | 3 | 2

ADVERSE EVENTS:
Time Frame: From study entry to end of study. The duration of follow up for a given participant was between 6 and 10 months depending on time of enrollment.
Description: From day 0-28, all SAEs, solicited AEs, and unsolicited AEs, with the exception of the following if not treated with prescription medication or over the counter medications with antipyretic properties: diaper rashes, teething pain, and spitting up. SAEs and LRIs were reported according to DAIDS EAE Manual V2.0 (see References). From day 29-56, SAEs were collected. After day 56, from November 1st - March 31 of the following year, medically attended fever, LRI, URI and otitis media were collected.
Groups:
- Vaccine: Participants received a single dose of the RSV LID cp ΔM2-2 vaccine at study entry (Day 0).
  RSV LID cp ΔM2-2 Vaccine: 10^5 plaque-forming units (PFUs); administered as nose drops
Arm/Group | Vaccine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/6
Serious Adverse Events (participants affected / at risk) | 4/11 | 2/6
Other Adverse Events (participants affected / at risk) | 9/11 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vaccine (N=11) | Placebo (N=6)
Bronchiolitis (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0
Croup infectious (Infections and infestations) | 1 | 0
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Vaccine (N=11) | Placebo (N=6)
Teething (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1
Discomfort (General disorders) | 1 | 2
Pyrexia (General disorders) | 5 | 4
Conjunctivitis (Infections and infestations) | 2 | 0
Conjunctivitis bacterial (Infections and infestations) | 1 | 0
Otitis media (Infections and infestations) | 1 | 0
Otitis media acute (Infections and infestations) | 5 | 0
Purulent discharge (Infections and infestations) | 1 | 0
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 1 | 0
Irritability (Psychiatric disorders) | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 4
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 6 | 6
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Stridor (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-08-08): https://cdn.clinicaltrials.gov/large-docs/81/NCT02890381/Prot_001.pdf
  • Statistical Analysis Plan (2016-09-02): https://cdn.clinicaltrials.gov/large-docs/81/NCT02890381/SAP_000.pdf